CLINICAL TRIAL: NCT05457153
Title: Intervention Protocol: Evaluation of the Effectiveness of the Technology-Based Well-Being Process Program (WEBEPROP) for Children and Adolescents in Palliative Care: A Randomized Trial
Brief Title: Technology-Based Well-Being Process Program (WEBEPROP) for Children and Adolescents in Palliative Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ebru Kilicarslan Toruner, Professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021 - 846
Record Dates: First submitted 2022-06-22; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Childhood Cancer
Keywords: Palliative Care; Spiritualitiy; Spiritual Care; Cancer; Child
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology-Based Well-Being Process Program (Experimental): WEBEPROP will be conducted for 8 weeks. The program for the intervention group is included the modüls. In the program, the modules of "Self-Knowledge, Inner Communication and Awareness of Perceptions, Emotion and Thought Management" will be completed in 8 weeks (each model two weeks) . The other module will not be accessible and cannot be switched before the prevous module is completed.
  Interventions: Other: Well-Being Process Program (WEBEPROP)
- Control Group (Active Comparator): After the first follow-ups have been made to the control group, they will continue to receive standard care. After the monitoring of the initiative group within the scope of the program is completed, the website of the well-being process program will be made available to the control group. Children and adolescents will benefit from the modules by promoting the website.
  Interventions: Other: Well-Being Process Program (WEBEPROP)

INTERVENTIONS:
Other: Well-Being Process Program (WEBEPROP) — Technology-Based Well-Being Process Program (WEBEPROP)

SUMMARY:
Objective: The research was planned to evaluate the effectiveness of the 8-week technology-based Well-Being Process program for children and adolescents in the palliative care period. Methods: This study was planned as a randomized controlled experimental study. The research will be carried out with children aged 12-20 years with a diagnosis of cancer, in the pediatric oncology and hematology clinics of two hospitals in Turkey. Data collection will consist of the children and adolescent's and parents' descriptive characteristic form Adolescent Spiritual Well-Being Scale, Beck Anxiety Scale, Pediatric Cancer Coping Scale and Technology-Based Spiritual Care Program Process Evaluation Forms. The program will be implemented for the intervention group. In the 8-week program; a) 4 web-based modules, b) 8 online individual interviews after each module (8 total interviews with each child) c) simultaneous mobile messages with the modules, and d) 24/7 counseling. Animation videos, breathing and progressive relaxation exercises, and imagination methods will be included in the modules. This research is based on the "Watson Model of Human Care".

DETAILED DESCRIPTION:
Hypothesis:

H1: There is a significant difference between the spiritual well being score averages of children and adolescents who have been administered and have not been administered WEBEPROP.

H2: There is a significant difference between the anxiety scores of children and adolescents who have been administered and have not been administered WEBEPROP.

H3: There is a significant difference between the coping scores of children and adolescents who have been administered and have not been administered WEBEPROP.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 10-20,
* Child and adolescent with palliative care needs
* At least 3 months before diagnosis
* Child and adoescent have completed the induction phase of treatment,
* İntermediate-high-risk group defined under a treatment protocol,
* Child and aolescent can utilizecomputer, mobile phone and tablet
* Children and adolescents who agreed to participate in the survey and their parent.

Exclusion Criteria:

* Newly diagnosed with physical and mental disabilities,
* Child and adolescent with severe anxiety according to the anxiety score scale,
* Out of diagnosis in the last 6 months (loss of parents, natural disaster, etc.) are children and adolescents who experience high levels of stress and have an important psychiatric diagnosis that affects their mental health.

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
The Scale of Spiritual Well-Being in Adolescents (SSWA) | The Scale of Spiritual Well-Beingscores will be checked at the beginning of the program "baseline"
  The scale developed by Törüner et al. assesses the spiritual well-being of adolescents aged 14-18 years. The scale, which is thought to help health professionals provide holistic care for adolescents, consists of a total of 34 items. Adolescents receive a minimum of 0 and a maximum of 136 points from the scale. As the score obtained from the scale increases, the spiritual well-being scores of adolescents increase. As the score obtained from the scale decreases, the spiritual well-being of the adolescents decreases. The Cronbach alpha value of the scale is 90.
Beck Anxiety Scale | Anxiety scores will be checked at the beginning of the program "baselıne
  The scale, which was developed by Beck et al. in 1988 to determine the level of anxiety (anxiety) of adult and adolescent individuals, consists of 21 items of the four-likert type. The Turkish validity and reliability study of the scale was conducted by Ulusoy et al. in 1993. Individuals are expected to be marked by their intensity of experiencing substances that are composed of symptoms and emotions commonly associated with anxiety. The sum of the scores was evaluated as 0-7: Minimal level of anxiety, 8-15: Mild level of anxiety, 16-25: Moderate level of anxiety, 26-63: Severe level of anxiety
Pediatric Cancer Coping Scale (PCCS) | Coping scores will be checked at the beginning of the program "baseline"
  The scale developed by Wu et al. for children with cancer between the ages of 7 and 18 years. The Turkish validity and reliability of the scale was conducted by Sengul and Törüner (2019). There are a total of 33 items in the scale. There are three sub-dimensions of cognitive coping, problem-oriented coping and defensive coping. A minimum of 0 and a maximum of 99 points is obtained from the scale. High scores obtained from the scale indicate high levels of coping strategies. A low score means that coping skills are insufficient.In the original study of the scale, the Cronbach Alpha value was determined as 0.91

SECONDARY OUTCOMES:
The Scale of Spiritual Well-Being in Adolescents (SSWA) | The Scale of Spiritual Well-Being scores will be checked completed"through study completion, an average of 1 week"
  The scale developed by Törüner et al. assesses the spiritual well-being of adolescents aged 14-18 years. The scale, which is thought to help health professionals provide holistic care for adolescents, consists of a total of 34 items. Adolescents receive a minimum of 0 and a maximum of 136 points from the scale. As the score obtained from the scale increases, the spiritual well-being scores of adolescents increase. As the score obtained from the scale decreases, the spiritual well-being of the adolescents decreases. The Cronbach alpha value of the scale is 90.
Beck Anxiety Scale | Anxiety scores will be checked completed"through study completion, an average of 1 week"
  The scale, which was developed by Beck et al. in 1988 to determine the level of anxiety (anxiety) of adult and adolescent individuals, consists of 21 items of the four-likert type. The Turkish validity and reliability study of the scale was conducted by Ulusoy et al. in 1993. Individuals are expected to be marked by their intensity of experiencing substances that are composed of symptoms and emotions commonly associated with anxiety. The sum of the scores was evaluated as 0-7: Minimal level of anxiety, 8-15: Mild level of anxiety, 16-25: Moderate level of anxiety, 26-63: Severe level of anxiety
Pediatric Cancer Coping Scale (PCCS) | Coping scores will be checked completed "through study completion, an average of 1 week"
  The scale developed by Wu et al. for children with cancer between the ages of 7 and 18 years. The Turkish validity and reliability of the scale was conducted by Sengul and Törüner (2019). There are a total of 33 items in the scale. There are three sub-dimensions of cognitive coping, problem-oriented coping and defensive coping. A minimum of 0 and a maximum of 99 points is obtained from the scale. High scores obtained from the scale indicate high levels of coping strategies. A low score means that coping skills are insufficient. In the original study of the scale, the Cronbach Alpha value was determined as 0.91

OTHER OUTCOMES:
The Scale of Spiritual Well-Being in Adolescents (SSWA) | The Scale of Spiritual Well-Beingscores will be checked completed, "through study completion, one month"
  The scale developed by Törüner et al. assesses the spiritual well-being of adolescents aged 14-18 years. The scale, which is thought to help health professionals provide holistic care for adolescents, consists of a total of 34 items. Adolescents receive a minimum of 0 and a maximum of 136 points from the scale. As the score obtained from the scale increases, the spiritual well-being scores of adolescents increase. As the score obtained from the scale decreases, the spiritual well-being of the adolescents decreases. The Cronbach alpha value of the scale is 90.
Beck Anxiety Scale | Anxiety scores will be checked completed, "through study completion, one month"
  The scale, which was developed by Beck et al. in 1988 to determine the level of anxiety (anxiety) of adult and adolescent individuals, consists of 21 items of the four-likert type. The Turkish validity and reliability study of the scale was conducted by Ulusoy et al. in 1993. Individuals are expected to be marked by their intensity of experiencing substances that are composed of symptoms and emotions commonly associated with anxiety. The sum of the scores was evaluated as 0-7: Minimal level of anxiety, 8-15: Mild level of anxiety, 16-25: Moderate level of anxiety, 26-63: Severe level of anxiety
Pediatric Cancer Coping Scale (PCCS) | Coping scores will be checked completed, "through study completion, one month
  The scale developed by Wu et al. for children with cancer between the ages of 7 and 18 years. The Turkish validity and reliability of the scale was conducted by Sengul and Törüner (2019). There are a total of 33 items in the scale. There are three sub-dimensions of cognitive coping, problem-oriented coping and defensive coping. A minimum of 0 and a maximum of 99 points is obtained from the scale. High scores obtained from the scale indicate high levels of coping strategies. A low score means that coping skills are insufficient. In the original study of the scale, the Cronbach Alpha value was determined as 0.91